CLINICAL TRIAL: NCT05632601
Title: Reexamining Her Cardiovascular Risk - Ottawa WomeN's Longitudinal Cohort Study
Acronym: HER-CROWN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20220586-01H
Record Dates: First submitted 2022-10-26; First posted 2022-11-30 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-07

CONDITIONS: Cardiovascular Diseases
Keywords: cardiovascular disease; sex-specific risk factor; hypertensive disorder of pregnancy; Early menopause; Polycystic ovarian syndrome; Rheumatologic inflammatory disorders; breast cancer; gestational diabetes; Primary ovarian insufficiency
MeSH Terms: conditions — Cardiovascular Diseases; Toxemia; Primary Ovarian Insufficiency; Polycystic Ovary Syndrome; Breast Neoplasms; Diabetes, Gestational | interventions — Positron-Emission Tomography

STUDY DESIGN:
Intervention Model Description: A single-site, two-group, matched-cohort Vanguard study will be completed to test feasibility outcomes to inform a large, multi-site, two-group, longitudinal matched-cohort study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sex-Specific Risk HDP Subgroup Factor Group and Age-Matched Control Group (Experimental): * Blood sample
  * Questionnaires
  * Arterial stiffness assessment
  * Transthoracic Echocardiogram
  * Coronary Computed Tomography Angiography (CTA)
  * Cardiac Positron Emission Tomography (PET)
  Interventions: Diagnostic Test: PET scan
- Sex-Specific Risk factor group and Age-Matched Control Group (No Intervention): * Blood sample
  * Questionnaires
  * Arterial stiffness assessment

INTERVENTIONS:
Diagnostic Test: PET scan — PET scan
  Arms: Sex-Specific Risk HDP Subgroup Factor Group and Age-Matched Control Group

SUMMARY:
The full HER CROWN will be a prospective cohort study to propose a novel, women-specific cardiovascular risk score/ algorithm in the prediction of hard cardiovascular outcomes (myocardial infarction, unstable angina, coronary revascularization, stroke, total and cardiovascular mortality). This future study will be the first longitudinal cohort study, to our knowledge, that is focused entirely on researching the pathophysiology and natural history of cardiovascular disease in women with known female-specific risk factors. Further, the investigators are aiming to recruit a sample that is representative of the ethnic distribution in Canada. The proposed pilot study is a feasibility study as an essential preparatory step for HER CROWN.

DETAILED DESCRIPTION:
Cardiovascular diseases (CVD), including ischemic heart disease (IHD), peripheral vascular disease (PVD), and stroke, remain the leading preventable cause of death among Canadian women, resulting in over 34,000 deaths per year (age-standardized death rate: 25.1%). Nearly 40% of CVD-related deaths in women are due to IHD. Increased awareness efforts and effective treatments have led to an overall decline in CVD mortality among men and women in high income countries over the past few decades; however, alarmingly, an increase in CVD mortality has been observed in women in the most recent 5 to 10 years in Canada and the United States, and an upward trend in rates of AMI among younger women.

CVD in women remains understudied, under-diagnosed, and undertreated. Clinical guidelines are largely based on studies of men. Several existing large longitudinal cohort studies (e.g., the Nurses' Health Study, The Framingham Heart Study, the PURE study) have included women; however, they have not focused recruitment specifically on high-risk cohorts of women or on risk factors that are unique to women, more common in women, or that disproportionately affect women; they have not used novel measures of subclinical disease in women (e.g., coronary computed tomography angiography and cardiac Rb-positive emission tomography); and most have not recruited representative samples of women in terms of ethnicity or socioeconomic status. CVD risk calculators (e.g., Framingham, the American College of Cardiology ASCVD) focus on traditional risk factors (e.g., tobacco smoking, hypertension, diabetes), do not include sex-specific CVD risk factors or factors that disproportionately affect women, and thus tend to underestimate risk in women. Female-specific factors that have been associated with CVD risk include: premature or late menarche, abnormal menses, premature or early menopause, gestational hypertensive disorders, gestational diabetes, preterm delivery, pregnancy loss, hormonal contraceptive use, and polycystic ovarian syndrome. Risk factors that are under-recognized or disproportionately affect women include: rheumatologic inflammatory disorders (RIDs), depression, anxiety, chronic stress, abuse and intimate partner violence, and health literacy. In addition, a more feminine gender role has been shown to be associated with higher risk of reinfarction after premature acute coronary syndrome, but no additional research on gender roles and future cardiovascular risk is available. Importantly, novel cardiovascular risk markers such as measures of arterial stiffness and aging, among others, have not been prospectively evaluated in a female population. As such, additional longitudinal research is needed to understand the natural history of CVD and the impact of these 'non-conventional' risk factors in women.

A recent article published in the Lancet by a multi-national group of women's heart health experts reviewed existing evidence, identified knowledge gaps, and provided specific recommendations related to CVD research, prevention, treatment, and access to care for women. The HER CROWN longitudinal cohort study will respond to three important gaps identified in this review, specifically: 1) describe the pathophysiology and natural history of cardiovascular disease in women; 2) determine the impact of sex-specific, psychosocial, and socioeconomic risk factors on CVD in women; and, 3) improve CVD risk prediction/ risk stratification models for women. The Vanguard phase of the study will evaluate the feasibility of the full study being planned.

The full HER CROWN will be a prospective matched-cohort study to propose a novel, women-specific cardiovascular risk score/ algorithm in the prediction of hard cardiovascular outcomes (myocardial infarction, unstable angina, coronary revascularization, stroke, total and cardiovascular mortality). This future study will be the first longitudinal cohort study, to our knowledge, that is focused entirely on researching the pathophysiology and natural history of cardiovascular disease in women with known female-specific risk factors. Further, the investigators are aiming to recruit a sample that is representative of the ethnic distribution in Canada. The proposed pilot study is a feasibility study as an essential preparatory step for HER CROWN. The study will be cross-disciplinary, including investigators who specialize in the treatment of cardiovascular disease in women, epidemiology and administrative data, cardiovascular imaging, biomarker research, physical activity, nutrition, nicotine addiction, and mental health who will each inform outcomes and sub-studies.

ELIGIBILITY:
Inclusion Criteria:

* Female Sex
* Between 25-55 years of age
* Ontario resident with a valid OHIP card

A prior or current diagnosis of:

* Pre-eclampsia, eclampsia, gestational hypertension
* Gestational diabetes
* Primary ovarian insufficiency (menopause < age 40)
* Early menopause (menopause between ages 40-45)
* Polycystic ovarian syndrome (PCOS)
* Rheumatologic inflammatory disorders (Lupus, Rheumatoid Arthritis, Psoriatic Arthritis)
* Breast cancer

OR

No prior history of sex-specific or female-predominant risk factors outlined in the SSR group

Exclusion Criteria:

* Male sex
* Currently pregnant
* Prior diagnosis of any of the following:
* CVD including coronary heart disease, heart failure, congenital heart disease, stroke/transient ischemic attack, valvular heart disease, peripheral vascular disease, aortapathy, atrial fibrillation or flutter, other CVD
* Neurodegenerative disease known to affect the heart (e.g., muscular dystrophy)
* Untreated serious mental illness (e.g., untreated psychosis)

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female sex
Enrollment: 210 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Demographics questionnaire | 18 months
  Demographics and socioeconomic information
Medical History Questionnaire | 18 months
  Past, present medical history, medication, and women's health related information
General Anxiety Disorder-7 (GAD-7) | 18 months
  This is calculated by assigning scores of 0, 1, 2, and 3 to the response categories, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." GAD-7 total score for the seven items ranges from 0 to 21.
  0-4: minimal anxiety 5-9: mild anxiety 10-14: moderate anxiety 15-21: severe anxiety
Patient Health Questionnaire (PHQ)-9 | 18 months
  Several days = 1 More than half the days = 2 Nearly every day = 3
  1-4 Minimal depression 5-9 Mild depression 10-14 Moderate depression 15-19 Moderately severe depression 20-27 Severe depression
Perceived Stress Scale (PSS) | 18 months
  PSS scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to the four positively stated items (items 4, 5, 7, & 8) and then summing across all scale items. A short 4 item scale can be made from questions 2, 4, 5 and 10 of the PSS 10 item scale.
The Index of Spouse Abuse (ISA) | 18 months
  Both the ISA-P and ISA-NP scores range from 0 to 100 where a low score indicates the relative absence of abuse and the higher scores represent the presence of a greater degree or amount of abuse.
Childhood Trauma Questionnaire (CTQ) | 18 months
  Responses are measured on a 5-point Likert scale (1 = never true, 2 = rarely true, 3 = sometimes true, 4 = often true, 5 = very often true). Each subscale is represented by five questions with a score range from 5 to 25; scores fall into four categories: none to low trauma exposure, low to moderate trauma exposure, moderate to severe trauma exposure and severe to extreme trauma exposure for each scale.
PTSD Checklist-5 (PCL-5) | 18 months
  Respondents are asked to rate how bothered they have been by each of 20 items in the past month on a 5- point Likert scale ranging from 0-4. Items are summed to provide a total severity score (range = 0-80). 0 = Not at all 1 = A little bit 2 = Moderately 3 = Quite a bit 4 = Extremely
SF-12 | 18 months
  SF-12v2 items are scored so that a higher score indicates a better health state. For example, functioning items are scored so that a high score indicates better functioning, and the pain item is scored so that a high score indicates freedom from pain. After data entry, items are scored in three steps:
  1. item recoding for the four items that require recoding;
  2. computing scale scores by summing across items in the same scale (raw scale scores); and,
  3. transforming raw scale scores to a 0-100 scale (transformed scale scores).
Substance use questionnaire | 18 months
  Nicotine, alcohol, cannabis use measure questionnaire. No score.
International Physical Activity Questionnaire (IPAQ) | 18 months
  Scoring a HIGH level of physical activity on the IPAQ means your physical activity levels equate to approximately one hour of activity per day or more at least a moderate intensity activity level. Scoring a MODERATE level of physical activity on the IPAQ means you are doing some activity more than likely equivalent to half an hour of at least moderate intensity physical activity on most days. Scoring a LOW level of physical activity on the IPAQ means that you are not meeting any of the criteria for either MODERATE of HIGH levels of physical activity.
The Newest Vital Sign (NVS) | 18 months
  Score by giving 1 point for each correct answer (maximum 6 points). Score of 0-1 suggests high likelihood (50% or more) of limited literacy. Score of 2-3 indicates the possibility of limited literacy. Score of 4-6 almost always indicates adequate literacy.
Arterial tonometry | 18 months
  Arterial stiffness and arterial age
Coronary CTA | 18 months
  Coronary artery calcium, plaque presence and plaque characteristics
Cardiac PET | 18 months
  Coronary perfusion and microvascular function
Transthoracic echocardiography | 18 months
  Cardiac structure and function
Blood work | 18 months
  CBC, electrolytes, creatinine, fasting lipids, fasting glucose, HbA1c, hs-troponin, NT-proBNP, Lipoprotein (a), LH, FSH, estradiol, progesterone, additional sample for biobanking βhCG test for subsamples participating in PET and Coronary CTA
Satisfaction Questionnaire | 18 months
  participant satisfaction and acceptability questionnaire. No score.

CONTACTS AND LOCATIONS:
Overall Officials: Kerri-Anne Mullen, PhD, Principal Investigator — UOHI
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No